CLINICAL TRIAL: NCT02963259
Title: Prospective Evaluation Comparing the Effects of Constant Current Versus Constant Voltage in Deep Brain Stimulation Using Hybrid Systems
Brief Title: IPG Replacement Study (PREFERENCE-H)
Acronym: PREFERENCE-H
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10135
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
Keywords: SJM Infinity™; SJM Brio™; Implantable pulse generator (IPG) replacement; SJM-CIP-10135; Deep brain stimulation (DBS)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SJM Infinity™ DBS IPG or a SJM Brio™ DBS IPG system: Subjects will be implanted with SJM Infinity™ DBS IPG or a SJM Brio™ DBS IPG system
  Interventions: Device: SJM Infinity™ DBS IPG or SJM Brio™ DBS IPG system

INTERVENTIONS:
Device: SJM Infinity™ DBS IPG or SJM Brio™ DBS IPG system — Implanted Medtronic® IPG will be explanted and replaced by a SJM Infinity™ DBS IPG or a SJM Brio™ DBS IPG system

SUMMARY:
This post-marketing evaluation has been designed to consistently investigate the subject's preference when switching from a Medtronic® constant voltage or constant current device to a St Jude Medical Infinity™ or St Jude Medical Brio™ constant current system. As electrodes will not be re-positioned, differences in subject's preference are to be explained by the difference in shape of the delivered pulse or waveform between the two systems.

ELIGIBILITY:
Inclusion Criteria:

* Subject (and caregiver, if applicable) signed the approved Informed Consent;
* Subject is ≥ 18 and ≤ 74 years of age;
* Subject is bilaterally treated with deep brain stimulation (DBS) in the subthalamic nucleus (STN) using a constant voltage device (i.e. Soletra™, Itrel™, Kinetra™, ActivaPC™ or ActivaRC™ IPG) and is responding satisfactory to CV stimulation in the Investigator's opinion;
* In the physician's opinion, the subject is a suitable candidate for an IPG replacement with different stimulation paradigm;
* Subject needs and/or requests an IPG replacement within 12 months after consent and the current IPG has at least 2.6 V output left (i.e. approx. 30% of full battery capacity) at the time of subject enrollment;
* PD symptom onset is no longer than 20 years;
* Subject has a Hoehn & Yahr score <IV (on stim);
* Subject with a normal cognitive function (MMSE ≥25);
* Subject is fluent speaker (as judged by the investigator) of the language spoken in the country where the investigational site is located.

Exclusion Criteria:

* IPG battery has less than 30% battery life at the time of consent;
* Need to replace or reposition the leads or extensions during the IPG replacement procedure;
* Subject had >10 recurrent falls experienced in the 3 months prior to consent;
* Subject is unwilling to change to either a St Jude Medical Infinity™ or Brio™ DBS system for the IPG replacement;
* Subject is unable to attend the study visits.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have a diagnosis matching the approved indication and are being considered for an IPG replacement comprise the target population of this study. All subjects who meet the inclusion and none of the exclusion criteria and have signed an Ethics Committee (EC) or Institutional Review Board (IRB) approved informed consent will be considered enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Karst, Study Director — Abbott
Locations (14):
- United States (3):
  - Baptist Hospital of Miami, Kendall, Florida
  - Neuroscience Consultants, Miami, Florida
  - Albany Medical College at Albany Medical Ctr, Albany, New York
- Germany (3):
  - Praxis Dr. Oehlwein, Gera
  - Klinik am Tharandter Wald, Halsbrücke
  - Universitätsklinikum Leipzig AÖR, Leipzig
- Italy (8):
  - Az.Osp. Universitaria Ferrara, Ferrara, Cona
  - Fondazione "Ospedale San Camillo" I.R.C.C.S, Padua, Veneto
  - Ospedale Generale Regionale F. Miulli, Acquaviva delle Fonti
  - Ospedale dell'Angelo, Mestre
  - IRCCS Istituto Ortopedico Galeazzi, Milan
  - Fondazione Istituto Neurologico Nazionale C. Mondino, Pavia
  - Policlinico Universitario A. Gemelli, Roma
  - Azienda Ospedaliero-Universitaria S Maria della Misericordia, Udine

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled a total of 17 subjects in 5 centers across Europe and United States between 29 March 2017 and 3 December 2018. Of the 17 enrolled subjects, 16 subjects were evaluated at the baseline visit and 12 completed the 3- and 12-month visit.
Pre-assignment Details: Of the total 17 participants enrolled, 5 were withdrawn for the reasons listed and only 16 completed the baseline.
Period: Overall Study
Arm/Group | SJM Infinity™ DBS IPG or a SJM Brio™ DBS IPG System
Started | 17
Completed | 12
Not Completed | 5
Not completed — IPG Replacement not Done with Abbott Device | 2
Not completed — Subject Participation Terminated by Investigator | 1
Not completed — Death | 1
Not completed — Subject Did Not Meet Inclusion/Exclusion Criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | SJM Infinity™ DBS IPG or a SJM Brio™ DBS IPG System
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4
  Italy | 12
UPDRS Score [Mean (Standard Deviation); unit: units on a scale] — The UPDRS score collected at baseline is relevant because it presents patient's baseline motor severity.
  The modified UPDRS retains the four-scale structure with a reorganization of the various subscales. Score ranges from 0 to 260, with 0 indicating no disability and 260 indicating total disability.
  units on a scale
    UPDRS III on stimulation | 23.6 (16.1)
    UPDRS III off stimulation | 39.8 (18.24)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Who Indicate Preference on Constant Current Over Constant Voltage at the 3 Month Follow-up Visit.
Description: Proportion of subjects who preferred constant current device over constant voltage, tested against a performance goal (PG) of 50.0% at the 3-month follow-up visit.
Time Frame: 3 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: participants
Arm/Group | SJM Infinity™ DBS IPG or a SJM Brio™ DBS IPG System
Number analyzed (Participants) | 12
participants | 4

2. Secondary Outcome: Number of Events Per Patient-year of Follow-up
Description: Total number of safety events related to battery replacement surgical procedures for hybrid systems divided by total follow-up duration from IPG replacement visit to either 12M visit or withdrawal visit (patient-years).
Time Frame: 12 months after IPG replacement
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: events per patient-year
Arm/Group | SJM Infinity™ DBS IPG or a SJM Brio™ DBS IPG System
Number analyzed (Participants) | 12
events per patient-year | 0

3. Secondary Outcome: Incidence Rate
Description: Number of subjects who underwent IPG replacement and encountered safety events related to battery replacement surgical procedure for hybrid system divided by total subjects who underwent IPG replacement.
Time Frame: 12 months after IPG replacement
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: subjects
Arm/Group | SJM Infinity™ DBS IPG or a SJM Brio™ DBS IPG System
Number analyzed (Participants) | 13
subjects | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | SJM Infinity™ DBS IPG or a SJM Brio™ DBS IPG System
All-Cause Mortality (participants affected / at risk) | 1/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 1/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SJM Infinity™ DBS IPG or a SJM Brio™ DBS IPG System (N=17)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SJM Infinity™ DBS IPG or a SJM Brio™ DBS IPG System (N=17)
High Impedance in Contact (Product Issues) | 1
Worsening of Motor/Parkinson's Disease Symptoms - Akinesia (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT02963259/Prot_SAP_000.pdf